CLINICAL TRIAL: NCT07322978
Title: Incidence of Splanchnic Venous Thrombosis in Acute Pancreatitis and it's Correlation With Severity of Pancreatitis - a Prospective Observational Study
Brief Title: Incidence of Splanchnic Venous Thrombosis in Acute Pancreatitis and it's Correlation With Severity of Pancreatitis
Status: Recruiting | Type: Observational
Sponsor: Asian Institute of Gastroenterology, India (Other)
Responsible Party: Sponsor
Other Study IDs: SVT in AP-01
Record Dates: First submitted 2025-04-02; First posted 2026-01-07 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-02

CONDITIONS: Acute Pancreatitis
MeSH Terms: conditions — Pancreatitis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Acute pancreatitis (AP) is a common medical condition characterized by inflammation of the pancreas, affecting a significant portion of the population. With approximately one-third of patients experiencing notable morbidity due to local or systemic complications, the severity of the disease is underscored by the presence of acute peripancreatic fluid collections, acute necrotic collections, pseudocysts, and walled-off necrosis1. Notably, vascular complications, such as splanchnic vein thrombosis, further contribute to the increased morbidity and mortality associated with acute pancreatitis2. Splanchnic vein thrombosis encompasses thromboses in the splenic (SpVT), portal (PVT), and superior mesenteric veins (SMVT), either individually or in combination3. These complications are often incidentally discovered during imaging procedures conducted to assess potential complications4. Despite most cases being asymptomatic, fatal complications, including bowel ischemia, liver failure, portal hypertension, and life-threatening bleeding, have been documented, with the risk of splanchnic vein thrombosis escalating with the severity of pancreatitis

DETAILED DESCRIPTION:
Acute pancreatitis (AP) is a common medical condition characterized by inflammation of the pancreas, affecting a significant portion of the population. With approximately one-third of patients experiencing notable morbidity due to local or systemic complications, the severity of the disease is underscored by the presence of acute peripancreatic fluid collections, acute necrotic collections, pseudocysts, and walled-off necrosis1. Notably, vascular complications, such as splanchnic vein thrombosis, further contribute to the increased morbidity and mortality associated with acute pancreatitis2. Splanchnic vein thrombosis encompasses thromboses in the splenic (SpVT), portal (PVT), and superior mesenteric veins (SMVT), either individually or in combination3. These complications are often incidentally discovered during imaging procedures conducted to assess potential complications4. Despite most cases being asymptomatic, fatal complications, including bowel ischemia, liver failure, portal hypertension, and life-threatening bleeding, have been documented, with the risk of splanchnic vein thrombosis escalating with the severity of pancreatitis.

The intricate relationship between the pancreas and large mesenteric vessels, coupled with systemic inflammatory responses, hypovolemia, fluid shifts, and prothrombotic states, contributes to the development of splanchnic vein thrombosis in acute pancreatitis5. Early detection of these thrombotic events becomes imperative to mitigate long-term sequelae such as portal hypertension and chronic mesenteric ischemia6. Despite the critical importance of identifying splanchnic vein thrombosis in acute pancreatitis, there is a notable absence of standardized recommendations for initiating anticoagulation treatment in these cases5. The decision-making process is further complicated by the potential risk of bleeding associated with other vascular complications, such as bleeding into pseudocysts or pseudo-aneurysmal bleeds7. As a result, there is a pressing need for more comprehensive studies that delve into the risk factors, pathogenesis, therapeutic impacts, and outcome predictors associated with splanchnic vein thrombosis in the context of acute pancreatitis. These investigations will not only enhance our understanding of the condition but also inform the development of evidence-based guidelines for the management of splanchnic vein thrombosis in individuals with acute pancreatitis.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 18-85 years of age.
* Diagnosis of AP as per international consensus criteria.

Exclusion Criteria:

* Chronic pancreatitis.
* Established malignancy.
* Cirrhosis of liver or established portal hypertension.
* Pregnancy.

Ages: 18 Years to 85 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All in-patients with acute pancreatitis, getting admitted from emergency or OPD will be enrolled. Only when a study subject has given informed consent, clinical data will be recorded
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2025-02-27 (Actual); Primary Completion 2026-02-27 (Estimated); Study Completion 2026-02-27 (Estimated)

PRIMARY OUTCOMES:
Primary outcome | 1 year
  Detection of thrombus in splenic, superior mesenteric or portal vein.

SECONDARY OUTCOMES:
Secondary Outcome | 1 year
  Correlation of splanchnic venous thrombosis with severity of acute pancreatitis.
Secondary Outcome | 1 year
  Incidence of infected pancreatic necrosis/ peri-pancreatic fluid collections in patients with acute pancreatitis having SVT.
Secondary Outcome | 1 year
  Effect of drainage of peripancreatic fluid collections/ necrotic collections on status of thrombosis.
Secondary Outcome | 6 months
  Vessel recanalization on follow-up at 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- AIG Hospital, Hyderabad, Telangana, India